CLINICAL TRIAL: NCT00417443
Title: A Study of Effect of Epidural Clonidine on Postoperative Pain Relief, Hyperalgesia and Chronic Pain in Patients Undergoing Colorectal Surgery
Brief Title: Epidural Clonidine for Postoperative Hyperalgesia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPICLO2006
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2006-12

CONDITIONS: Postoperative Hyperalgesia
Keywords: epidural; clonidine; hyperalgesia; laparotomy
MeSH Terms: conditions — Hyperalgesia | interventions — Clonidine

INTERVENTIONS:
Drug: Clonidine

SUMMARY:
We propose performing a study in which we compare the effects of bupivacaine and fentanyl with a different drug combination - bupivacaine and clonidine. The principal research questions of the study are:

1. To compare the effect of clonidine (with bupivacaine), injected into the epidural space on the extent of hyperalgesia (abnormal pain/sensitivity in the uninjured skin surrounding the operation site) in patients undergoing operations for bowel disease, with that of fentanyl (with bupivacaine).
2. To compare the effect of clonidine (with bupivacaine), injected into the epidural space on the incidence of chronic pain 6 months after surgery for bowel disease, with that of fentanyl (with bupivacaine).

DETAILED DESCRIPTION:
In addition to pain at the surgical incision site, patients undergoing major bowel operations commonly experience pain in the surrounding (uninjured)skin during the postoperative period - this phenomenon is known as hyperalgesia. In most patients hyperalgesia resolves with healing of the wound, but in some patients it persists. Recent studies have shown that 25% of patients undergoing bowel surgery will have chronic pain at 1 year following surgery. This pain can be debilitating and has significant implications, both for the individual and for society. For the individual there are significant physical, mental, social and economic implications. The burden on society is significant because bowel surgery operations are very common, and many of the 25% of the patients who develop chronic pain will required ongoing treatment and unable to work.Chronic pain after surgery is believed to be a result of changes in the central nervous system (i.e. brain and spinal cord)occurring during and immediately after the surgery. Indeed the likelihood of a patient developing chronic pain is related to the extent of hyperalgesia during the initial post-operative period. Two other important predisposing factors are the emotional state of the patient and the genetic predisposition of the patient to develop chronic pain states. In our hospital, in common with most western hospitals, patients undergoing major bowel surgery commonly have an epidural catheter (a soft plastic tube inserted in the space surrounding the spinal cord fluid) inserted before the operation to facilitate the administration, during the first few postoperative days, of a combination of a local anaesthetic agent (bupivacaine in our hospital) and an opiate drug (a morphine-like medicine; fentanyl is used in our hospital). Unfortunately, neither fentanyl nor bupivacaine appear to reduce the incidence of hyperalgesia. In fact there is evidence that larger doses of opiates such as fentanyl can increase the extent and severity of hyperalgesia. Moreover, although routinely used in our hospital, fentanyl is associated with several adverse effects including nausea and vomiting, generalised itching, sedation (sleepiness), and respiratory depression (slowed respiration rate). Recent studies have shown that when clonidine is injected through an epidural catheter, it can provide good pain relief in the immediate post-operative period, and is also effective in reducing the extent of hyperalgesia in the area around the incision. This, in turn may lead reduce the probability of patients developing persistent pain. There is good evidence to show that when clonidine is used instead of fentanyl, the adverse effects are reduced.

Although epidural clonidine has been used with success in different surgical settings, there are no published studies comparing epidural combinations of bupivacaine and clonidine with bupivacaine and fentanyl (or all 3 drugs together) in patients undergoing abdominal surgery. There is now good evidence from animal and human studies to suggest that a combination of fentanyl and clonidine has more pain-relieving effect than either of the two drugs administered on its own.

We thus propose to compare the pain relieving effects of these three drug combinations in patients undergoing abdominal operations for bowel resection.

There are various methods of detecting hyperalgesia. Measurement of sensitivity to touch and pain in the skin around the incision site is a simple and reproducible method. This involves use of simple devices - a brush (to test pain on touch) and a plastic pointed hair/filament (to detect and measure abnormal sensitivity to a mildly painful stimulus in the area around the incision). To determine the incidence of chronic pain we will follow up patients after surgery by telephoning to ask them questions relating to the intensity of their pain as well as its effect on their lifestyle. To assess the patients' emotional state before surgery we will ask them to complete questionnaires known to be reliable and validated for detection of anxiety and depression, for assessment of general well-being. For detection of genetic predisposition to developing chronic pain, we will analyse patients' blood samples for genes that are known to either reduce the effectiveness of pain-relieving medication,or to make them more sensitive to painful stimuli.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years
2. Scheduled for elective major bowel surgery through a vertical midline incision
3. An epidural catheter for pain relief during and after the operation is required and the patient has already consented to it.
4. Good physical health or if they have any disease (e.g. heart disease, high blood pressure, asthma), it should be well controlled with medication.

Exclusion Criteria:

1. Previous abdominal surgery, kidney or liver disease
2. Inability to understand or comply with the study protocol
3. Allergy to any of the study drugs
4. Failure of either placement of an epidural catheter or poor pain relief with epidural analgesia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-12; Study Completion 2009-12

PRIMARY OUTCOMES:
Extent of peri-incisional hyperalgesia in patients undergoing laparotomy for bowel disease
Incidence of chronic pain 6 months after laparotomy for bowel disease

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Absalom, MBBS MD FRCA, Principal Investigator — Addenbrooke's NHS Trust, Cambridge, United Kingdom
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom